CLINICAL TRIAL: NCT04289779
Title: A Phase 2 Study of CAbozantinib in Combination with AtezolizumaB As NeoAdjuvant Treatment for Muscle-Invasive BladdEr Cancer
Brief Title: Study of CAbozantinib in Combination with AtezolizumaB for Muscle-Invasive BladdEr Cancer
Acronym: ABATE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Deepak Kilari (Other)
Collaborators: Exelixis (Industry); Genentech, Inc. (Industry); Medical College of Wisconsin (Other)
Responsible Party: Sponsor-Investigator, Deepak Kilari, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU18-343
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Bladder Cancer
Keywords: muscle invasive
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — cabozantinib; atezolizumab; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Cabozantinib 40 mg orally daily x 9 weeks plus Atezolizumab 1200 mg every 3 weeks x 3 doses
  Interventions: Drug: Cabozantinib; Drug: Atezolizumab; Procedure: Cystectomy

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib 40 mg orally daily for 3 cycles
  Other Names: cabometyx
Drug: Atezolizumab — Atezolizumab 1200 mg IV every 3 weeks for 3 cycles
  Other Names: Tecentriq
Procedure: Cystectomy — Patients will receive three cycles of treatment prior to cystectomy unless they discontinue treatment for unacceptable toxicity or progressive disease by RECIST v1.1 or withdraw consent.

SUMMARY:
This is an open-label phase II study assessing the activity of cabozantinib combined with atezolizumab in patients with resectable muscle-invasive urothelial carcinoma who are ineligible for cisplatin-based therapy or decline cisplatin-based therapy. Each cycle equals 21 days. The dose of atezolizumab is 1200 mg IV flat dose every 3 weeks (Day 1) plus cabozantinib 40 mg orally daily (Day 1 through Day 21). Patients will receive three cycles of treatment prior to cystectomy unless they discontinue treatment for unacceptable toxicity or progressive disease by RECIST v1.1 or withdraw consent.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥18 years at the time of consent.
* ECOG Performance Status of ≤ 2 within 28 days prior to registration.
* Histological or cytologically confirmed muscle-invasive urothelial carcinoma of the bladder. Urothelial carcinoma invading into the prostatic stroma with no histologic muscle-invasion is allowed.
* Archival tissue is required, if available. The tissue should be identified at screening and shipped after registration, prior to Cycle 3 Day 1. If archival tissue is not available a repeat biopsy is not required, and the subject may still be eligible. Archival tissue should have been obtained within 60 days prior to registration.
* Urothelial carcinoma should be the predominant component (≥ 50%). NOTE: Any neuroendocrine differentiation is not permitted.
* Clinical stage T2-T4aN0/xM0 disease.
* No clinical or radiographic evidence for locally advanced or metastatic disease.
* Medically appropriate candidate for radical cystectomy as assessed by surgeon.
* Patients must have a contraindication to cisplatin or decline cisplatin based neoadjuvant chemotherapy. Absolute or relative contraindication to cisplatin, defined as one or more of the following within 28 days prior to registration (Grading per CTCAE v5):

  * Creatinine clearance < 60 mL/min (Cockcroft-Gault formula will be used to calculate creatinine clearance)
  * Grade ≥ 2 hearing loss
  * Grade ≥ 2 neuropathy
* No radiation therapy < 4 weeks of registration. NOTE: prior radiation therapy to the bladder is not allowed.
* Recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatment.
* Must have a life expectancy of at least 12 weeks at registration.
* Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 28 days prior to registration. See protocol for more details.

  * White blood cell count ≥ 2500/mm3 (≥2.5 GI/L)
  * Absolute Neutrophil Count (ANC) ≥ 1500/mm3 (≥1.5 GI/L) without G-CSF
  * Platelet Count (Plt) ≥ 100,000/mm3 (≥100 GI/L) without transfusion
  * Hemoglobin (Hgb) ≥ 9 g/dL (may be transfused)
  * Calculated creatinine clearance ≥ 30 mL/min per Cockcroft-Gault formula
  * Urine protein/creatinine ratio (UPCR) ≤ 2 mg/mg if no hematuria and ≤ 3.5 mg/mg if hematuria noted
  * Calcium or ionized calcium; Calcium <12 mg/dL or corrected serum calcium < ULN or ionized calcium <1.5 mmol/L
  * Bilirubin ≤ 1.5 × upper limit of normal (ULN); if documented Gilbert's syndrome bilirubin must be ≤ 3 x ULN
  * Albumin ≥ 2.8 g/dl.
  * Aspartate aminotransferase (AST) ≤ 2.5 × ULN
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN
  * Alkaline Phosphatase ≤ 2.5 x ULN
  * International Normalized Ratio (INR) or Prothrombin Time (PT); Activated Partial Thromboplastin Time (aPTT) ≤ 1.3 × ULN (Applies only to subjects not receiving therapeutic anticoagulation; subjects receiving therapeutic anticoagulation should be on a stable dose)
* No radiation therapy < 4 weeks of registration. NOTE: prior radiation therapy to the bladder is not allowed.
* Recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatment.
* Must have a life expectancy of at least 12 weeks at registration.
* Negative HIV test at screening; NOTE: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥200/µL, and have an undetectable viral load.
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. The HBV DNA test will be performed only for patients who have a positive total HBcAb test.
* Negative total hepatitis C core antibody (HCcAb) test at screening, or positive total HCcAb test followed by a negative hepatitis C virus (HCV) DNA test at screening. The HCV DNA test will be performed only for patients who have a positive total HCcAb test.
* Females of childbearing potential must have a negative urine or serum pregnancy test within 30 days prior to registration. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* Females of childbearing potential and males must be willing to abstain from heterosexual intercourse or to use 2 forms of effective methods of contraception from the time of informed consent (females) or initiation of treatment (males) until 5 months (150 days) after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method. Males should not donate sperm and women should not breastfeed or store breast milk for the timeframe outlined above.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Prior treatment with cabozantinib.
* Severe infection within 4 weeks prior to initiation of study treatment per investigator assessment. Examples include hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety.
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Active infection requiring systemic therapy.
* Active tuberculosis.
* Prior history of stem cell or solid organ transplantation.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during the study or within 5 months after the last dose of study drug.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Treatment with any investigational drug within 30 days prior to registration.
* Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or other cancer for which the subject has been disease-free for at least five years. Patients with localized prostate cancer who are either being followed by an active surveillance program OR planning to undergo definitive treatment are also eligible.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins. NOTE: Previously identified allergy or hypersensitivity to components of the study treatment formulations or history of severe infusion-related reactions to monoclonal antibodies are excluded. Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption are also excluded.
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab or cabozantinib formulation.
* Prior treatment with the following is prohibited unless otherwise specified:

  * Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies or systemic chemotherapy (prior intravesical induction immunotherapy for non-muscle invasive disease is allowed).
  * Any type of small molecule kinase inhibitor within 2 weeks before first dose of study treatment.
  * Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy within 4 weeks before first dose of study treatment.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest imaging.
* Significant cardiovascular disease, such as:

  * New York Heart Association Congestive Heart Failure Class II or greater.
  * Myocardial infarction, unstable angina or unstable arrhythmias within 3 months of enrollment.
  * History of stroke or TIA within 3 months of enrollment.
  * Other clinically significant arterial vascular disease within 6 months of enrollment (e.g. aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis). Prior history of adequately treated venous thromboembolism > 7 days prior to C1D1 on stable dose of therapeutic anticoagulation is permitted.
  * Subjects with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed.
* History of leptomeningeal disease.
* Uncontrolled tumor-related pain. Patients requiring pain medication must be on a stable regimen at study entry.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.

Atezolizumab-Specific Exclusion Criteria

* Treatment with systemic immunostimulatory agents (including but not limited to IFNs, interleukin [IL]-2) within 6 weeks or five half-lives of the drug, whichever is shorter, prior to Cycle 1 Day 1.
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1 Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial (Subjects who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled ).The use of inhaled corticosteroids, physiologic replacement doses of glucocorticoids (i.e., for adrenal insufficiency), and mineralocorticoids (e.g., fludrocortisone for adrenal insufficiency) is allowed. The use of prednisone 10 mg or equivalent dose of steroids is also allowed.
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, granulomatosis with polyangiitis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Exceptions include:

  * Subjects with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
  * Graves' disease.
  * Subjects with controlled Type I diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
  * Subjects with a history of celiac disease may be eligible if controlled with diet.
  * Skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment.
  * Conditions not expected to recur in the absence of an external trigger.

Cabozantinib -Specific Exclusion Criteria

* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  --Cardiovascular disorders:
  * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
  * History of additional risk factors for torsades de pointes (e.g., long QT syndrome)
* Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

  * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
  * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. NOTE: Complete healing of an intra-abdominal abscess must be confirmed before first dose.
  * Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
* Hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose.
* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
* Lesions invading or encasing any major blood vessels.
* Other clinically significant disorders that would preclude safe study participation.

  * Serious non-healing wound/ulcer/bone fracture.
  * Uncompensated/symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
* Major surgery (eg, GI surgery) within 2 weeks before C1D1. Complete wound healing from major surgery and from minor surgery (eg, simple excision, tooth extraction) must have occurred prior to treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* For subjects with known QTcF of > 500 ms, corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment. NOTE: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Concomitant anticoagulation with coumarin agents (eg, warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (eg, clopidogrel). Allowed anticoagulants are the following:

  * Low-dose aspirin for cardioprotection (per local applicable guidelines) is permitted.
  * Low-dose low molecular weight heparins (LMWH) are permitted. Prophylactic use of anticoagulants is allowed.
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* Uncontrolled gross hematuria associated with clots per investigator's discretion.
* Inability to swallow pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic Response Rate | 12 months
  Estimate the pathologic response (PaR) rate to neoadjuvant cabozantinib and atezolizumab in subjects with muscle-invasive urothelial cancer of the bladder. Pathologic response rate (PaR) is defined as the absence of residual muscle-invasive cancer in the surgical specimen (pathologic downstaging to ≤ pT1pN0), which includes pT0, pT1, pTa, and pTis

SECONDARY OUTCOMES:
Frequency and Severity of Adverse Events | 12 months
  Assess the frequency and severity of adverse events per CTCAE v5
Pathologic complete response rate | 12 months
  Estimate the pathologic complete response (pCR) rate to neoadjuvant cabozantinib and atezolizumab in subjects with muscle-invasive urothelial cancer of the bladder. pCR rate is defined as the proportion of patients whose pathological staging was T0N0M0 as assessed per local institutional pathology review using specimens obtained via cystectomy following the neoadjuvant treatment.
Event Free Survival | 24 months
  EFS is defined as the time from registration to the first recurrence of disease after cystectomy, the time of first documented progression in patients who are precluded from cystectomy, or the time of death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Kilari, MD, Principal Investigator — Medical College of Wisconsin
Locations (6):
- United States (6):
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No